CLINICAL TRIAL: NCT04623931
Title: Phase II Trial of Treatment Intensification for IDH Wildtype, Non-Histological Glioblastoma, Gliomas (IDH Wildtype Lower Grade Glioma Treatment Intensification)
Brief Title: Chemotherapy and Radiation Therapy for the Treatment of IDH Wildtype Gliomas or Non-histological (Molecular) Glioblastomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0715; NCI-2019-08264 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0715 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-05-19; First posted 2020-11-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Anaplastic Astrocytoma, IDH-Wildtype; Anaplastic Oligoastrocytoma; Anaplastic Oligodendroglioma; Diffuse Astrocytoma, IDH-Wildtype; Glioblastoma; Oligoastrocytoma; Oligodendroglioma; WHO Grade II Glioma; WHO Grade III Glioma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma | interventions — Radiotherapy; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (temozolomide, radiation therapy) (Experimental): Patients receive temozolomide PO daily and radiation therapy over 5 days a week (weekdays only) for 6 weeks. Beginning 28 days after the last dose of radiation therapy, patients receive temozolomide PO for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Temozolomide

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase II trial studies how well temozolomide and radiation therapy work in treating patients with IDH wildtype historically lower grade gliomas or non-histological molecular glioblastomas. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving chemotherapy with radiation therapy may kill more tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. The goal of this clinical research study is to compare receiving new radiation therapy doses and volumes to the prior standard treatment for patients with historically grade II or grade III IDH wild-type gliomas, which may now be referred to as IDH wildtype molecular glioblastomas at some institutions. Receiving temozolomide in combination with radiation therapy may also help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the progression free survival (PFS) based on Response Assessment in Neuro-Oncology (RANO) imaging criteria from start of treatment with concurrent chemoradiation (CRT) and adjuvant temozolomide (TMZ).

SECONDARY OBJECTIVE:

I. To determine the 3-year overall survival (OS) of isocitrate dehydrogenase (IDH) wild-type grade II and grade III gliomas with dose escalation radiation with concurrent chemoradiation therapy.

EXPLORATORY OBJECTIVES:

I. To assess local control patterns (site of 1st progression). II. To evaluate neuro-cognitive function by the Neurocognitive Clinical Trial Battery (CTB).

III. To evaluate the treatment related symptoms, overall symptom impact, and disease related factor groupings utilizing the M.D. Anderson Symptom Inventory Brain Tumor (MDASI-BT).

IV. To assess the quality of life.

OUTLINE:

Patients receive temozolomide orally (PO) daily and radiation therapy over 5 days a week (weekdays only) for 6 weeks. Beginning 28 days after the last dose of radiation therapy, patients receive temozolomide PO for 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1, 3, 5, 7, 9, 12, 15, 18, 21, 24, 28, 32, and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Historical grade II and III gliomas IDH wildtype gliomas by including; diffuse astrocytoma, anaplastic astrocytoma, oligodendroglioma, anaplastic oligodendroglioma, oligoastrocytoma, anaplastic oligoastrocytoma
* IDH wildtype gliomas (molecularly defined high grade glioma or molecularly defined glioblastoma [GBM])
* History & physical exam, and Karnofsky performance status (KFS) of >= 70 within 30 days prior to enrollment
* Post-operative magnetic resonance imaging (MRI) with contrast is mandatory and necessary for radiation therapy (RT) planning
* Thin-slice (< 1.5 mm) three-dimensional (3D) T1 pre and post contrast and axial T2/fluid-attenuated inversion recovery (FLAIR) sequences for planning purposes are highly encouraged to obtain.
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (within 60 days prior to registration)
* Platelets >= 100,000 cells/mm^3 (within 60 days prior to registration)
* Hemoglobin >= 10.0 g/dl (within 60 days prior to registration) (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 10.0 g/dl is acceptable)
* Bilirubin =< 1.5 upper limit of normal (ULN) (within 60 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (within 60 days prior to registration)
* Blood urea nitrogen (BUN) < 30 mg/dl (within 60 days prior to registration)
* Serum creatinine < 1.5 mg/dl (within 60 days prior to registration)

Exclusion Criteria:

* Definitive clinical or radiologic evidence of metastatic disease; if applicable
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years. (For example, carcinoma in situ of the breast, oral cavity or cervix are permissible)
* Prior cranial radiotherapy or radiotherapy to the head and neck where potential field overlaps would exist
* Prior chemotherapy or radiotherapy for any brain tumor
* Histologic diagnosis of gliosarcoma World Health Organization (WHO grade IV) or pilocytic astrocytoma (WHO grade I)
* Multicentric glioblastoma
* Leptomeningeal disease
* Inability to undergo MRI with and without contrast
* Severe, active co-morbidity defined as follows:

  * Unstable angina or congestive heart failure requiring hospitalization within 6 months prior to enrollment
  * Transmural myocardial infarction within the last 6 months prior to registration. Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of >= 2 mm using the analysis of an electrocardiogram (EKG) performed within 28 days prior to registration. (Note: EKG to be performed only if clinical suspicion of cardiac issue)

    • New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to registration
  * Serious and inadequately controlled arrhythmia at step 2 registration
  * Serious or non-healing wound, ulcer or bone fracture or history of abdominal fistula, intra-abdominal abscess requiring major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to registration, with the exception of the craniotomy for surgical resection
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for coagulation parameters are not required for entry into this protocol
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Human immunodeficiency virus (HIV) positive with CD4 count < 200 cells/microliter. Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is because the treatments involved in this protocol may be significantly immunosuppressive with potentially fatal outcomes in patients already immunosuppressed
* Any other severe immunocompromised condition
* Active connective tissue disorders, such as lupus or scleroderma that in the opinion of the treating physician may put the patient at high risk for radiation toxicity
* End-stage renal disease (i.e., on dialysis or dialysis has been recommended)
* Any other major medical illnesses or psychiatric treatments that in the investigator's opinion will prevent administration or completion of protocol therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From start of treatment until objective tumor progression or death, whichever happens first, assessed up to 52 months
  Tumor progression is defined by the Response Assessment in Neuro-Oncology glioma criteria. PFS time will be estimated using the Kaplan-Meier method. The 1-year PFS rate will be estimated along with a 95% confidence interval. Patient or tumor characteristics (ex. grade, age, etc) will be compared within the single study cohort. Cox regression models will be applied to assess the effect of covariates of interest on PFS.

SECONDARY OUTCOMES:
Overall survival (OS) rate | From start of treatment until death from any cause, assessed at 3 years
  The 3-year OS rate is defined as the proportion of participants that are alive at 3-year after the start of treatment, which will be estimated along a 95% confidence interval. OS time will be estimated using the Kaplan-Meier method. Patient or tumor characteristics (ex. grade, age, etc) will be compared within the single study cohort. Cox regression models will be applied to assess the effect of covariates of interest on OS.

OTHER OUTCOMES:
Local control patterns (site of 1st progression) | Up to 3 years
  Will be summarized with frequency and proportion.
Neuro-cognitive function | Up to 3 years
  Assessed by the Neurocognitive Clinical Trial Battery, and summarized with descriptive summary statistics.
Symptom burden | Up to 3 years
  Assessed by the M.D. Anderson Symptom Inventory Brain Tumor (MDASI-BT), and summarized using standard descriptive statistics such as mean, standard deviation, median and range. Wilcoxon rank-sum test or Kruskal Wallis test will be used to examine the difference on MDASI-BT between or among patients' characteristics groups.
Quality of life | Up to 3 years
  Assessed by linear analog self-assessment (LASA) scale, will be summarized using standard descriptive statistics such as mean, standard deviation, median and range. Wilcoxon rank-sum test or Kruskal-Wallis test will be used to examine the difference on LASA scale between or among patients' characteristics groups.

CONTACTS AND LOCATIONS:
Overall Officials: Debra N Yeboa, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org